CLINICAL TRIAL: NCT04356131
Title: The Effect of Massage and Progressive Relaxation Exercises on Pain Intensity and Menstrual Symptoms of Students With Primary Dysmenorrhoea
Brief Title: Effect of Massage and Progressive Relaxation Exercises on Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, EBRU YILDIZ, Principal Investigator, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: pain management
Record Dates: First submitted 2020-04-16; First posted 2020-04-22 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Primary Dysmenorrhea
Keywords: Dysmenorrhoea; Massage; Progressive relaxation exercises; Pain; Menstrual symptom; Randomized controlled trial
MeSH Terms: conditions — Dysmenorrhea; Pain | interventions — Massage

STUDY DESIGN:
Intervention Model Description: The study was done experimentally in pre-test and post-test design and randomized controlled model among students with PD.
  The sample size was calculated with power analysis. According to calculations, it was found that 58 students were enough for sampling through 95% of power value, 0.05 of confidence interval and 0.88 of effect size. Students who were determined to meet sampling and inclusion criteria through questionnaire and accepted to participate in the study were assigned into the experimental and control groups through randomization.
  During the follow-up of the three menstruation periods, the number of groups was increased in case of drop-out and 100 students were included. However, the study was completed with a total of 97 students -50 students for the experimental group and 47 students for the control group- because 3 students of the control group withdrew from the study in the second month.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Students in the experimental group were taught about massage and progressive relaxation exercises (PRE). The phases of the massage and PRE trainings were first explained by being demonstrated by the author on herself. In the meantime, the trainings were video-taped and uploaded to the mobile phones of the students. After the author, each student was made to perform massage and PRE. Both the exercises and massage techniques were daily performed 3 times a day after pain had started and relaxation exercises lasted 30 minutes whereas massage was performed for 15 minutes consecutively
  Interventions: Other: progressive relaxation exercises and massage
- control group (No Intervention): The students in the control group continued their routines during the study.

INTERVENTIONS:
Other: progressive relaxation exercises and massage — Progressive relaxation exercises included 30 minute rhythmic breathing and muscle relaxation exercises were demonstrated in the second part of the CD with river sounds and verbal instructions. Massage techniques were performed on the site between upper symphysis pubis and umbilicus with 15 minute effleurage demonstrated in the third part of the CD with nature sound.
  Arms: experimental group

SUMMARY:
A total of 97 female students, 50 in the intervention group and 47 in the control group, were included in this pretest-posttest design randomized controlled study. Massage and progressive relaxation exercises are self-administered practices that are easy to adopt, with no side effects, and have beneficial effects on pain, sweating, fatigue, and gastrointestinal and central nervous system signs. So, it can be asserted that when applied together, massage and progressive relaxation exercises could be more effective in reducing menstrual symptoms than applying them separately.

DETAILED DESCRIPTION:
Dysmenorrhea is one of the most frequent problems during menstruation and described as periodic and painful pelvis menstruation among women at reproductive age. It is classified as primary and secondary dysmenorrhea. Primary dysmenorrhea (PD) is defined as suprapubic pelvis pain with cramps that begin a couple hours before menstrual bleeding, after menstrual bleeding, or during the last 12-72 hours of menstruation and occur repeatedly without organic pathology. PD is associated with an increase in prostaglandin production in the endometrium, which causes pain by increasing uterine contractions in the suprapubic region. According to De Sanctis et al., PD prevalence varies between 16% and 93%. It is often seen with sweating, fatigue, gastrointestinal system signs (lack of appetite, nausea, vomiting, diarrhea), and central nervous system signs (dizziness, headache, syncope, and lack of concentration). These symptoms that occur just before or just after menstrual bleeding among women with normal pelvic anatomy may prevent them from attending school and work or joining social activities. Secondary dysmenorrhea is defined as menstrual pain caused by a pathology in the pelvis such as endometriosis. If a patient has pain for 3-6 months, a more comprehensive evaluation of chronic pelvic pain should be performed to evaluate the potential etiologies of secondary dysmenorrhea.

The international literature includes oral contraceptive, nonsteroidal anti-inflammatory, and sedative drugs for the treatment of primary dysmenorrhea. However, the fact that some of these drugs cause side effects such as indigestion, headache, drowsiness, and substance addiction causes individuals to remain indifferent to them. In Turkey, it is reported that women prefer their family members as the first source of information and therefore use individual methods (massage, herbal teas, hot application, lying down, sweet food consumption, etc.) rather than pharmacological treatments due to cultural differences in coping with PD. Complementary and integrated therapy approaches, which are widely used all over the world today, have become common in coping with gynecological disorders among women in recent years. Some studies state that PD can be cured using such complementary therapies as essential oil acids, vitamins, acupuncture, herbal medicines, aromatherapy, reflexology, acupressure, massage, sports, and exercise. However, ACOG emphasizes that although these methods are frequently used by patients, they have not been studied enough yet, and mostly supports the use of exercise, high-frequency transcutaneous electrical nerve stimulation, and topical heat to help manage dysmenorrhea symptoms. Research on PD has applied massage and exercise practices using different application protocols. Studies on massage applications have examined the effect of inhaling herbal essential oils alone or together with massage. Research solely on exercise has examined the effectiveness of long-term and regular exercise, although with various practices. However, it can be said that massage and progressive relaxation exercises are more advantageous than other methods because they are easy, economical, and can be applied without the need for someone else.

Massage intensifies the blood flow in the area of application and reduces muscle tension. It also increases endorphin secretion and raises the pain threshold. Relaxation exercises, on the other hand, provide a decrease in sympathetic activity, an increase in parasympathetic activity and consequently a widening of the peripheral vessels, an increase in blood flow in the blood vessels, and a decrease in muscle tension and pain perception. Moreover, it has been reported that pain, anxiety, and depression symptoms decrease as a result of the decrease in the activation of the sympathetic nervous system, thanks to the deep breathing exercises performed during PRE. Therefore, it is predicted that massage combined with PRE will be beneficial in PD management. In this sense, this study was conducted to examine the effect of massage and PRE together on pain severity and other menstrual symptoms in PD treatment.

The literature includes no studies on the use of massage and PRE together in PD management. Therefore, the aim of the current study was to examine the effect of massage and PRE together on pain intensity and other menstrual symptoms in the management of PD.

ELIGIBILITY:
Inclusion Criteria:

* Being older than 18 years,
* Having a dysmenorrhea pain intensity score ≥4 according to Visual Analog Scale (VAS),
* Having no previous pregnancy experience,
* Having no disease that leads to dysmenorrhea,
* Using no hormonal contraception or intrauterine device,
* Having a menstruation period of 3-8 days and a menstrual cycle of 21-35 days,
* Having no systemic-chronic disease or physical/mental health problems that prevent/restrict massage or exercise,
* Volunteering to participate in the study.

Exclusion Criteria:

* Being younger than 18 years
* Having a dysmenorrhea pain intensity score ≤ 4 according to Visual Analog Scale (VAS),
* Having previous pregnancy experience,
* Having disease that leads to dysmenorrhoea (endometriosis, ovarian cysts/tumors, pelvic infection disease, myoma/uterus tumor, uterus polyp, asherman syndrome, infection),
* Using hormonal contraception and intrauterine devices,
* Not to present a menstruation period that lasts 3-8 days and menstrual cycle of 21-35 days,
* Having a systemic and chronic disease (diabetes, heart diseases, vein diseases, circulatory disorders, varicosis, blood diseases, etc.),
* Having any physical/mental health problems that prevent/restrict massaging and exercising,
* Not to be voluntary to join the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Primary dysmenorrhoea is described as painful menstrual periods among women who have normal pelvic anatomy and causes physical and psychological health to be affected with hormonal changes as well as some symptoms such as nausea, vomiting, fatigue and stress.
Enrollment: 97 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Students' individual and menstruation-related characteristics as assessed by "The Personal Information Form". | 1 day
  At the pretest stage of the research, by the experimental group and control group, "The Personal Information Form" form is filled in to specify individual characteristics and menstruation period characteristics.

SECONDARY OUTCOMES:
Students' Menstruation Period Pain as assessed by The short-form McGill Pain Questionnaire. | 28 day
  By the experimental group in each menstrual period for 3 consecutive months: both the exercises and massage techniques were daily performed three times a day after pain had started and relaxation exercises lasted 30 minutes whereas massage was performed for 15 minutes and after that the form is filled in.
  Without any application by the control group the form is filled in after pain start.
  In the form, pain quality is determined with 15 descriptors that describe sensory (first 11) and affective pain (last 4). Dimension of pain is evaluated to demonstrate the intensity by using a rating of 0-3 (0=none, 1=mild, 2=moderate, 3=severe). Pain quality scores of sensory pain (0-33 score), of affective pain (0-12 score) and of total (0- 45 score) are obtained. A rise in total pain quality score indicates a rise in pain sensory. In the study in order to provide an overall intensity score; Visual analog scale is included in the scale. Visual analog scale suggests general pain intensity.
Students' Menstruation Period Menstrual Symptoms as assessed by Daily Symptom Rating Scale. | 28 day
  By the experimental group in each menstrual period for 3 consecutive months: both the exercises and massage techniques were daily performed three times a day after pain had started and relaxation exercises lasted 30 minutes whereas massage was performed for 15 minutes and after that "Daily Symptom Rating Scale" form is filled in.
  Without any application by the control group "Daily Symptom Rating Scale" form is filled in after menstrual symptoms start.
  In the scale that includes 17 symptoms, each symptom is scored according to its intensity with a five point rating between 0 and 5. An increase in scores indicates high intensity of the symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University Faculty of Nursing, Mersin, Turkey (Türkiye)

REFERENCES:
- [Background] Avcı D.K, Sarı E. Approach to dysmenorrhea and effect of dysmenorrhea on social life and school performance in the university students. Van Medical Journal. 2018; 25(2): 188-193.
- [Background] Azima S, Bakhshayesh H.R, Mousavi S, Ashrafizaveh S. Comparison of the effects of reflexology and massage therapy on primary dysmenorrhea. Biomedical Research. 2015; 26 (3): 0976-1683.
- [Background] De Sanctis V, Soliman A, Bernasconi S, Bianchin L, Bona G, Bozzola M, Buzi F, De Sanctis C, Tonini G, Rigon F, Perissinotto E. Primary Dysmenorrhea in Adolescents: Prevalence, Impact and Recent Knowledge. Pediatr Endocrinol Rev. 2015 Dec;13(2):512-20. PMID 26841639
- [Background] Memmott J. The effect of music-assisted progressive muscle relaxation on the self-reported symptoms of women with primary dysmenorrhoea [PhD thesis]. Kansas: University of Kansas; 2009.
- [Background] Apay SE, Arslan S, Akpinar RB, Celebioglu A. Effect of aromatherapy massage on dysmenorrhea in Turkish students. Pain Manag Nurs. 2012 Dec;13(4):236-40. doi: 10.1016/j.pmn.2010.04.002. Epub 2010 Sep 15. PMID 23158705
- [Background] İbrahimoğlu Ö, Kanan N. The effect of progressive muscle relaxation exercises after endotracheal extubation on vital signs and anxiety level in open heart surgery patients. Turk Journal Intense Care. 2017; 15(3): 98-106.
- [Background] Mackereth PA, Booth K, Hillier VF, Caress AL. Reflexology and progressive muscle relaxation training for people with multiple sclerosis: a crossover trial. Complement Ther Clin Pract. 2009 Feb;15(1):14-21. doi: 10.1016/j.ctcp.2008.07.002. Epub 2008 Oct 1. PMID 19161949